CLINICAL TRIAL: NCT01772784
Title: Effects of Phenolic Acids on Endothelial Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 11.36.NRC
Record Dates: First submitted 2012-07-25; First posted 2013-01-21 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2012-11

CONDITIONS: Healthy
Keywords: subjects

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- phenolic acids (Experimental): Maltodextrine + Phenolic acids
  Interventions: Other: Phenolic acids
- placebo (Placebo Comparator): Maltodextrine
  Interventions: Other: Phenolic acids
- phenolic acid (Experimental): Maltodextrine + Phenolic acids
  Interventions: Other: Phenolic acids
- polyphenol (Active Comparator)
  Interventions: Other: Phenolic acids

INTERVENTIONS:
Other: Phenolic acids — Phenolic acids

SUMMARY:
Epidemiological studies suggest dietary (poly) phenols decrease the risk of death from cardiovascular diseases. (Poly)phenol-rich foods include fruits and vegetables as well as tea, coffee, red wine, and chocolate. The aim of the present study is to investigate whether endothelial function is altered by ingestion of phenolic acids. Moreover, the investigators will evaluate the effect of phenolic acids on blood pressure and platelet adhesion.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* males
* Smokers

Exclusion Criteria:

Any food allergy

* Abnormal blood pressure defined as follow: systolic <100 or >160 mmHg and diastolic <50 or >100mmHg
* Regular consumption of medication within 2 months before the study inclusion
* Caffeine intake 1 day before screening measurements (and 1 day before each visit),
* Any intake of multivitamin-tablets and other supplemental compounds 10 days before the study start and throughout the study.
* Excessive alcohol intake defined as > 280 g per week

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-06; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
endothelial dysfunction | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Yves Allemann, MD, Prof., Principal Investigator — University Hospital, Bern, Switzerland
Locations (1):
- Swiss Cardiovascular Center Bern, University Hospital, Bern, Switzerland

REFERENCES:
- [Derived] Mills CE, Flury A, Marmet C, Poquet L, Rimoldi SF, Sartori C, Rexhaj E, Brenner R, Allemann Y, Zimmermann D, Gibson GR, Mottram DS, Oruna-Concha MJ, Actis-Goretta L, Spencer JPE. Mediation of coffee-induced improvements in human vascular function by chlorogenic acids and its metabolites: Two randomized, controlled, crossover intervention trials. Clin Nutr. 2017 Dec;36(6):1520-1529. doi: 10.1016/j.clnu.2016.11.013. Epub 2016 Nov 30. PMID 28012692